CLINICAL TRIAL: NCT02422472
Title: Comparison of Ultrasound Guided Peripheral IV Placement With and Without Use of a Guidewire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Heidi Kimberly, Associate Physician Emergency Medicine Brigham and Women's Hospital, Instructor in Emergency Medicine Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015P000073
Record Dates: First submitted 2015-04-14; First posted 2015-04-21 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Difficult Peripheral IV Access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (No Intervention): Standard of care ultrasound guided peripheral IV placement
- Experimental (Experimental): Ultrasound guided peripheral IV placement with the use of a guidewire
  Interventions: Device: Ultrasound guided peripheral IV placement

INTERVENTIONS:
Device: Ultrasound guided peripheral IV placement — Accucath™ 20 Gax 5.7cm catheter
  Arms: Experimental

SUMMARY:
The purpose of this study is to compare ultrasound guided peripheral IV placement with and without the use of a guidewire. Patients in the Emergency Department with difficult peripheral IV access (as defined by 2 failed attempts by nursing staff) will be consented and randomized to standard ultrasound guided peripheral IV placement or ultrasound guided peripheral IV placement with modified seldinger technique using a guidewire.

ELIGIBILITY:
Inclusion Criteria:

* Difficult peripheral IV access (2 failed attempts by nursing staff)
* Prior history of difficult IV access and patient request for ultrasound guided IV

Exclusion Criteria:

* Need for emergent access or central venous access
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
First attempt success rate | 60 minutes
  First attempt success is defined as ability to place and use the catheter after only one attempt and will be reported by study staff.

SECONDARY OUTCOMES:
Overall success rate | 60 minutes
  Overall success is defined as ability to place and use the catheter (after 2 or fewer attempts) and will be reported by study staff.
Number of skin punctures | 60 minutes
  Number of skin punctures will be recorded by study staff.
Complications including hematoma, IV infiltration, catheter dislodge | 3 days
  Patients will be monitored for complications of IV placement by study staff

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Kimberly, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No